CLINICAL TRIAL: NCT01417806
Title: A Phase II Trial of SOM230(PasireotideLAR) and Topotecan in Patients With Relapsed or Refractory Small Cell Lung Cancer
Brief Title: Trial of pasireotideLAR and Topotecan in Relapsed or Refractory Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Florida Veterans Affairs Foundation for Research and Education (U.S. Federal Agency)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Niramol Savaraj, M.D. Lucy Chua M.D. Vy Dinh M.D. Medhi Wangpaichits PhD, VA. Medical Center, Miami, Fl
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230DUS21T
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-07

CONDITIONS: Small Cell Lung Cancer
Keywords: small cell lung cancer; somatostatin; topotecan
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan; pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Topotecan and Pasireotide — Topotecan 1.5mg/m2 dailyx5 days and Pasireotide 60 mg IM every 28 days

SUMMARY:
The majority of small cell lung cancer(SCLC)(50-100%) express somatostatin receptors(type 1-5) with some small cell lung cancer express more than one subtypes. Stimulation of these SSTR's lead to inhibition of angiogenesis and cell growth. SOM230 also lower levels of IGF which is known to contribute to SCLC proliferation. Topotecan is approved for second line therapy in relapsed small cell lung cancer. We hypothesized that combination of both agents should yield greater antitumor activity.

DETAILED DESCRIPTION:
The primary objectives of this study is to assess the progression-free survival (PFS) with the combination of SOM230 and topotecan in patients with SCLC who relapsed or progressed after front-line chemotherapy with cisplatin and etoposide. The secondary objective is to evaluate the efficacy and safety of SOM230 in combination with topotecan in this population. The primary end point is progression free survival. The secondary objective is response rate duration of response , overall survival , safety and tolerability. Patient who is eligible for the study will received topotecan 1.5mg/m2 on day 1-5 and SOM230 60mg on day 1 every 28 days until tumor progression or toxicity limit further treatment. Contrast-enhanced CT scans will be performed at baseline and every 2 months (or sooner if clinically indicated) to assess the response, duration of response, and time to tumor progression Patients will be allowed to remain on therapy if treatment is tolerated and if there is no evidence of progression for a maximum of 1 year or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion criteria

1. Histologically documented SCLC failed one chemotherapy with documentation of relapse or progressive disease.
2. Measurable or evaluable disease by CT scan. If evaluable disease or measurable disease has been previously treated, this must show signs of tumor progression by CT.
3. Karnofsky performance status of 80, Age ≥ 18 years and life expectancy of ≥12 weeks
4. Minimum of four weeks since any major surgery, completion of radiation or chemotherapy
5. ANC ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hgb > 9 g/dL.
6. Serum bilirubin ≤ 2 x upper limit of normal (ULN), and serum transaminases activity ≤ 3 x ULN, with the exception of serum transaminases (< 5 x ULN) if the patient has liver metastases. Serum creatinine ≤ 1.5 x ULN.
7. Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: If exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
8. Women of childbearing potential must have a negative serum pregnancy test within 14 days of the administration of the first study treatment. Women must not be lactating.
9. Signed informed consent to participate in the study must be obtained from patients after they have been fully informed of the nature and potential risks by the investigator (or his/her designee) with the aid of written information.

Exclusion criteria

1. Prior topotecan or prior octreotide therapy.
2. Chronic treatment with systemic steroids or another immunosuppressive agent.
3. Patients should not receive immunization with attenuated live vaccines during study period or within 1 week of study entry.
4. Uncontrolled brain or leptomeningeal metastases.
5. Patients with prior or concurrent malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, or other cancer from which the patient has been disease free for five years.
6. Patients with uncontrolled diabetes mellitus or a fasting plasma glucose > 1.5 ULN..
7. Patients with symptomatic cholelithiasis.
8. Patients who have congestive heart failure, unstable angina, sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia, advanced heart block or a history of acute myocardial infarction within the six months preceding enrollment.
9. Patients who are at high risk for cardiac arrhythmias as defined by any of the following:

   * Baseline QTcF > 450 msec
   * History of syncope or family history of idiopathic sudden death or long QT syndrome
   * Sustained or clinically significant cardiac arrhythmias
   * Risk factors for Torsades de Pointes such as hypokalemia, hypomagnesemia, cardiac failure, clinically significant/symptomatic bradycardia, or high-grade AV block
   * Concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by diabetes, or Parkinson's disease), HIV, cirrhosis, uncontrolled hypothyroidism or cardiac failure
   * Concomitant medication(s) known to increase the QT interval
10. Patients taking concomitant medications that are at risk of prolonging QT interval. If patient is to be included in the study, these medications need to be discontinued
11. Patients with the presence of active or suspected acute or chronic uncontrolled infection or with a history of immunocompromise, including a positive HIV test result
12. None malignant disease that are uncontrolled such as severe impaired lung function.
13. Women who are pregnant or breast feeding, or women/men able to conceive and unwilling to practice an effective method of birth control. (Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to administration of pasireotide). Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study.
14. Known hypersensitivity to somatostatin analogues or any component of the pasireotide or octreotide LAR formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2011-07; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 5 years
  Primary outcome Progression free survival (PFS).

SECONDARY OUTCOMES:
response rate and overall survival | 5 years
  Secondary outcome Response rate (RR), duration of response, overall survival (OS), safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Niramol Savaraj, M.D., Principal Investigator — VA.Medical Center Miami, Fl. 33125
Locations (1):
- VA. Medical Center, Miami, Florida, United States